CLINICAL TRIAL: NCT05581186
Title: Efficacy of Pulse Electromagnetic Field Therapy (PEMF) in Patients With Nonspecific Chronic Neck Pain: A Randomized Controlled Study
Brief Title: Efficacy of Pulse Electromagnetic Field Therapy (PEMF) in Patients With Nonspecific Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Nur Doğanlar, Medical research assistant, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NECKPEMF2022
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Neck Pain; Musculoskeletal Diseases; Chronic Neck Pain; Cervical Disc Disease
Keywords: Pulse Electromagnetic Field Therapy; Chronic neck pain; Cervical Disc Disease
MeSH Terms: conditions — Neck Pain; Musculoskeletal Diseases | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PEMT + exercise (Active Comparator): A total of 15 sessions of pulse electromagnetic field therapy using an electromagnetic field device (ASA Pmt Quatro Pro, ASA Srl Via A.Volta 9-36057, Italia),five times a week and once a day for three weeks, were applied to the patients. The patients were then given a daily exercise program once a day by a physiotherapist.
  Interventions: Other: Pulse electromagnetic field therapy
- Sham PEMT + exercise (Sham Comparator): Sham therapy was applied in five sessions a week for three weeks, with a total of 15 sessions, with no current flowing through the device. This was followed by the exercise programs described above, performed once a day with the physiotherapist.
  Interventions: Other: Sham pulse electromagnetic field therapy
- Exercise only (Other): Exercise program was applied in five sessions a week for three weeks, with a total of 15 sessions a day with the physiotherapist.
  Interventions: Other: Therapeutic Exercise

INTERVENTIONS:
Other: Pulse electromagnetic field therapy — It was applied with an electromagnetic field device (ASA Pmt Quatro Pro, ASA Srl Via A.Volta 9-36057 Italia) at 25 Hz frequency, 30 Gauss, %35 intensity and for 25 minutes. The treatment period was 5 days a week for 3 weeks, in total. It was applied as 15 sessions.
  Therapeutic Exercise As a therapeutic exercise program (neck stability exercises); active cervical ROM, cervical isometric and progressive (selfexercise with Thera-Band) strengthening muscles; trapezius, scalene, rhomboid, levator scapular, pectoral, suboccipital muscles stretching exercises, scapular stabilization exercises. It was planned to implement a total of 15 sessions 5 days a week for 3 weeks, for approximately 30 minutes. Exercises will be performed by a trained (at least 5 years experienced) physiotherapist, three times a day, in 3 sets, 10 repetitions.
  Arms: PEMT + exercise
Other: Sham pulse electromagnetic field therapy — Sham pulse electromagnetic field therapy was applied five sessions a week for four weeks, for a total of 15 sessions a day, using electromagnetic field device (ASA Pmt Quatro Pro, ASA Srl Via A.Volta 9-36057 Italy) without current flowing through the device.
  Therapeutic Exercise As a therapeutic exercise program (neck stability exercises); active cervical ROM, cervical isometric and progressive (selfexercise with Thera-Band) strengthening muscles; trapezius, scalene, rhomboid, levator scapular, pectoral, suboccipital muscles stretching exercises, scapular stabilization exercises. It was planned to implement a total of 15 sessions 5 days a week for 3 weeks, for approximately 30 minutes. Exercises will be performed by a trained (at least 5 years experienced) physiotherapist, three times a day, in 3 sets, 10 repetitions.
  Arms: Sham PEMT + exercise
Other: Therapeutic Exercise — Therapeutic Exercise As a therapeutic exercise program (neck stability exercises); active cervical ROM, cervical isometric and progressive (selfexercise with Thera-Band) strengthening muscles; trapezius, scalene, rhomboid, levator scapular, pectoral, suboccipital muscles stretching exercises, scapular stabilization exercises. It was planned to implement a total of 15 sessions 5 days a week for 3 weeks, for approximately 30 minutes. Exercises will be performed by a trained (at least 5 years experienced) physiotherapist, three times a day, in 3 sets, 10 repetitions.
  Arms: Exercise only

SUMMARY:
This investigation aims to investigate the effectiveness of Pulse Electromagnetic Field Therapy (PEMF) on neck pain, cervical range of motion, pressure pain threshold and quality of life in patients with nonspecific chronic neck pain compared to cervical therapeutic exercises.

DETAILED DESCRIPTION:
Neck pain is a common musculoskeletal complaint in society. It is the most common musculoskeletal problem after low back pain. It may regress spontaneously within a few weeks or may become chronic, as in 30% of patients. When it becomes chronic, it can negatively affect the daily life activities of individuals and lead to functional limitations and inadequacies.

Various approaches exist for neck pain in clinical practice. Among them; education of patients on neck pain, ergonomic arrangements, analgesics, non-steroidal anti-inflammatory drugs, muscle relaxants, exercise, physical therapy agents such as transcutaneous electrical stimulation (TENS), superficial and deep heaters, Pulse Electromagnetic Field Therapy (PEMT) , manipulation, mobilization methods, nerve blockages and surgical intervention.

Magnetotherapy is a treatment method based on magnetic field interaction. As a result of pulsed or alternating electromagnetic fields, an electrical current occurs in the tissues. Pulse magnetotherapy has three physical mechanisms known to be effective in living tissue: Magnetic induction, magneto-mechanical effects, and electronic interactions. Effects of magnetic field application are vasodilation, analgesic effect, anti-inflammatory effect, acceleration of healing, antiedematous effect. Magnetotherapy increases the oxygen release of erythrocytes and provides oxygenation of the tissues. This causes a decrease in toxins in the damaged area, an increase in vital nutrients and endorphins. With this physiological change, magnetic energy decreases the pain receptor sensitivity that sends a message to the brain. With this treatment method, pain reduction is achieved, while joint mobility increases. This investigation was designed prospective sham controlled randomized study. Participants were randomized into 3 groups: PEMT + therapeutic exercise, sham PEMT + therapeutic exercise, and only therapeutic exercise. As evaluation parameters, cervical range of motion, Visual Pain Scale (VAS) Neck, Visual Pain Scale (VAS) Neck, SF (Short form) -36 Quality of Life Scale, pressure pain threshold measurement with an algometer, patient global assessment, and physician global assessment will be evaluated with.It was planned that the evaluations were made and recorded by a blinded physician to the groups at the beginning of the treatment, at the end of the treatment and at the 6th week controls.

ELIGIBILITY:
Inclusion Criteria:

1. Neck pain for at least 3 months in the 20-55 age range
2. Diagnosed with nonspecific chronic neck pain by examination, history and imaging methods

Exclusion Criteria:

1. Pregnancy
2. Inflammatory rheumatologic diseases
3. Malignity
4. Having a cardiac pacemaker
5. Previous surgery related to the cervical spine
6. Having bleeding diathesis
7. Having a body implant with an electronic or battery system
8. Neck pain due to neurological and vascular diseases
9. Having neurological diseases
10. Having received physical therapy and rehabilitation for the cervical area in the last 6 months
11. Acute infections

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline visual analog scale (VAS) neck and arm pain at 3rd and 6th week | up to 6th week
  Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity.

SECONDARY OUTCOMES:
Change from baseline quality of life (short form 36 (SF-36)) at 3rd and 6th weeks | up to 6th week
  This is a self-administered scale, which is widely used to measure the quality of life. It was developed to measure the quality of life in patients who have physical illnesses; however, it can also be successfully used in healthy individuals and patients who have psychiatric diseases. SF-36 includes 36 items and surveys eight domains of health, such as physical functionality, physical role limitations, pain, general health, vitality, social functionality, emotional role limitations, and mental health. Total score was between 0 ( disability) and 100 (no disability). Every subgroup of the questionnaire has a score scale between 0 and 100. Every increase in the subgroup of SF-36 questionnaire, which is a positive scoring system, indicates increase in quality of life related to health.
Change from baseline range of motion of cervical spine measurements with goniometer at 3rd and 6th weeks | up to 6th week
  Cervical flexion, extension ,lateral flexion ,rotations(goniometric measurement results in units of degrees).
Change from baseline Neck Dısabılıty Index (NDI) at 3rd and 6th weeks | up to 6th week
  The Neck Disability Index (NDI) is designed to measure neck-specific disability. The questionnaire has 10 items concerning pain and activities of daily living including personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation. Each question measures from 0 to 5, the total score out of 100 is calculated.
Change from baseline Pressure pain threshold measurement with an algometer at 3rd and 6th weeks | up to 6th week
  The algometer is a useful tool for determining pressure pain threshold measurements. Pressure pain threshold is defined as the minimum force applied to elicit pain. A digital pressure algometer (Baseline, push-pull, force gauce Algometer, USA) will be used for measurements. The most painful point in the cervical region will be determined by sitting all patients in their most comfortable position for measurement. Three measurements will be made at an angle of 90 to this point, repeated at 1-minute intervals, and the average of these three measurements will be taken and this value will be recorded as the mean pressure pain threshold in kg/cm2. During the measurement, the value at the first moment when the patient feels pain will be taken as a basis.
Change from baseline In the global evaluation of the patient at 3rd and 6th weeks | up to 6th week
  "Very bad" is written on the end corresponding to the numerical value of "0 cm" and "very good" is written on the end corresponding to the numerical value of "10 cm".
Change from baseline In the doctor's global evaluation at 3rd and 6th weeks | up to 6th week
  "Very bad" is written on the end corresponding to the numerical value of "0 cm" and "very good" is written on the end corresponding to the numerical value of "10 cm".

CONTACTS AND LOCATIONS:
Locations (1):
- Nur Doğanlar, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dusunceli Y, Ozturk C, Atamaz F, Hepguler S, Durmaz B. Efficacy of neck stabilization exercises for neck pain: a randomized controlled study. J Rehabil Med. 2009 Jul;41(8):626-31. doi: 10.2340/16501977-0392. PMID 19565156
- [Background] Griffiths C, Dziedzic K, Waterfield J, Sim J. Effectiveness of specific neck stabilization exercises or a general neck exercise program for chronic neck disorders: a randomized controlled trial. J Rheumatol. 2009 Feb;36(2):390-7. doi: 10.3899/jrheum.080376. PMID 19132780
- [Background] Karakas M, Gok H. Effectiveness of pulsed electromagnetic field therapy on pain, functional status, and quality of life in patients with chronic non-specific neck pain: A prospective, randomized-controlled study. Turk J Phys Med Rehabil. 2020 May 18;66(2):140-146. doi: 10.5606/tftrd.2020.5169. eCollection 2020 Jun. PMID 32760890
- [Background] Sutbeyaz ST, Sezer N, Koseoglu BF. The effect of pulsed electromagnetic fields in the treatment of cervical osteoarthritis: a randomized, double-blind, sham-controlled trial. Rheumatol Int. 2006 Feb;26(4):320-4. doi: 10.1007/s00296-005-0600-3. Epub 2005 Jun 29. PMID 15986086
- [Background] Hattapoglu E, Batmaz I, Dilek B, Karakoc M, Em S, Cevik R. Efficiency of pulsed electromagnetic fields on pain, disability, anxiety, depression, and quality of life in patients with cervical disc herniation: a randomized controlled study. Turk J Med Sci. 2019 Aug 8;49(4):1095-1101. doi: 10.3906/sag-1901-65. PMID 31385489